CLINICAL TRIAL: NCT06280001
Title: A Multicenter Prospective Clinical Cohort Study on the Pathogen Spectrum of HIV/AIDS Complicated With Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Beijing Ditan Hospital (Other); Beijing YouAn Hospital (Other); Huashan Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jiajia Chen, Chief Physician of the First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang University
Other Study IDs: 2023YFC2308802-04
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: Infection; Pathogen spectrum; Cohort study
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — According to the characteristics of infection, take blood or body fluids from the corresponding infected site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine the incidence and spectrum of opportunistic infections among Chinese HIV/AIDS patients at this stage, to find intervention targets, to construct an early warning prediction model, and to give an individualized program with integrated immune function to obtain salvage opportunities for patients.The main questions it aims to answer are:

* Describe the populations and characteristics of pathogenic microorganisms involved in HIV co-infection, map the spatial and temporal changes in the infection system of pathogenic microorganisms, and evaluate their impact on disease regression.
* Explore the mechanism of interaction between pathogenic microorganisms and host autoimmune deficiencies.
* Discover early warning and predictive markers and immunological indicators of pathogenic microorganisms, and explore new technologies and programs to reduce the mortality rate of infection.

DETAILED DESCRIPTION:
AIDS is a chronic systemic disease caused by human immunodeficiency virus (HIV), which leads to reduced or defective immune function, causing a variety of serious opportunistic infections and tumors, and a significant increase in the mortality rate. This study focuses on the impact of secondary infections on the clinical prognosis of patients with HIV/AIDS, and intends to establish a prospective, multicenter clinical cohort of HIV/AIDS patients with combined infections with a variety of pathogens, to map the infectious pathogens, to correlate the characteristics of the basic immune status with the spectrum of pathogens of secondary infections, and to establish a monitoring and early-warning system of secondary infections, so that we can explore safe and effective treatments to further reduce the disease and mortality rate.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form.
2. HIV positive.
3. Any gender, age 18 to 70 years old

Exclusion Criteria:

1.Patients deemed unsuitable by the investigator to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/AIDS patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Secondary infections in patients with HIV/AIDS at 4 weeks | 4 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or Next-generation sequencing(NGS) results.
quick SEPSIS RELATED ORGAN FAILURE ASSESSMENT(qSOFA) at 4 weeks | 4 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.

SECONDARY OUTCOMES:
Survival rate | 12 weeks
  12-week survival in patients with HIV/AIDS co-infection with secondary infections.

CONTACTS AND LOCATIONS:
Overall Officials: Jiajia Chen, Principal Investigator — Zhejiang University